CLINICAL TRIAL: NCT00345215
Title: The Effect of High and Low Sodium Intake on Aquaporin-2 in Healthy Humans, During Basal Conditions and After Hypertonic Saline Infusion.
Brief Title: The Effect of High and Low Sodium Intake on Urinary Aquaporin-2 in Healthy Humans.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Responsible Party: Carolina Cannillo Graffe, Department of Medical Research, Holstebro Hospital
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: med.res.hos.2006.cc.01
Record Dates: First submitted 2006-06-24; First posted 2006-06-27 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Healthy Humans
Keywords: Urinary Aquaporin 2; High/low Sodium Diet; Fractional Sodium Excretion
MeSH Terms: interventions — Diet, Sodium-Restricted

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: High Sodium Diet — 250-350 mmol
Behavioral: Low Sodium Diet — 25-35 mmol

SUMMARY:
The aim of the study is to test the hypothesis that the function and/or regulation of aquaporin 2 and/or endothelial sodium channels in the principal cells of healthy humans is abnormal at high and low sodium intake

ELIGIBILITY:
Inclusion Criteria:

* Caucasic men and women
* Age 18-65 years
* Body mass index less or equal to 30 Kg/m2

Exclusion Criteria:

* Arterial hypertension
* History or clinical signs of heart, brain, lung, kidney, malignant or endocrine organ disease.
* Abnormal biochemical screening of the blood regarding: red and white cell count, B-hemoglobin, P-sodium, P-potassium, P-creatinine, P-albumine, P- bilirubin, P-alanine aminotransferase, P- alkaline phosphatase, p-cholesterol and B-glucose.
* Abnormal screening of the urine regarding: blood, albumine and glucose.
* Alcohol or drug abuse
* Drug use except oral contraceptives
* Smoking
* Abnormal electrocardiogram
* Blood donation within one month of the first examination day
* Pregnancy
* Unwillingness to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-05; Primary Completion 2006-12 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
u-AQP-2 | Before and after hypertonic saline infusion after 4 days on high and low sodium diet, respectively.
fractional sodium excretion | Before and after hypertonic saline infusion after 4 days on high and low sodium diet, respectively.
p-aldosterone | Before and after hypertonic saline infusion after 4 days on high and low sodium diet, respectively.

SECONDARY OUTCOMES:
u-pAQP-2 | Before and after hypertonic saline infusion after 4 days on high and low sodium diet, respectively.
u-ENaC(alfa-beta-gamma) | Before and after hypertonic saline infusion after 4 days on high and low sodium diet, respectively.
CH20 | Before and after hypertonic saline infusion after 4 days on high and low sodium diet, respectively.
ucAMP | Before and after hypertonic saline infusion after 4 days on high and low sodium diet, respectively.
uPGE2 | Before and after hypertonic saline infusion after 4 days on high and low sodium diet, respectively.
GFR | Before and after hypertonic saline infusion after 4 days on high and low sodium diet, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Erling B. Pedersen, Professor, Study Chair — Department of Medical Research, Holstebro Hospital, Denmark; Carolina C. Graffe, MD, Principal Investigator — Department of Medical Research, Holstebro Hospital, Denmark
Locations (1):
- Department of Medical Research, Holstebro Hospital, Holstebro, Holstebro, Denmark